CLINICAL TRIAL: NCT04091477
Title: Impact of Neuropsychological Alteration of Decision-making Abilities on the Functioning of Patients With Eating Disorders
Brief Title: Impact of Neuropsychological Alteration of Patients With Eating Disorders
Acronym: NeuropsyTCA
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: INSERM 1061-Montpellier (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0436
Record Dates: First submitted 2019-09-13; First posted 2019-09-16 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2019-09

CONDITIONS: Eating Disorder
Keywords: Anorexia nervosa; Bulimia; Binge eating disorders; Neuropsychology; neurocognition; Daily functioning
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia; Binge-Eating Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Eating disorders are multifactorial disorders currently conceptualized in a biopsychosocial model, but pathophysiology remains relatively unknown, and robust etiological models to guide treatment are therefore lacking. Different endophenotypes and neurocognitive vulnerability factors have been found in eating disorders including decision making abnormalities. The investigators hypothesize that decision making abnormalities are associated with a lower level of functioning and quality of life which could lead to social and interpersonal difficulties. The investigators also hypothesize that these anomalies are associated with a particular clinical profile (more restrictive profile, more hyperactivity, less insight on the disease and desire for care ...).

DETAILED DESCRIPTION:
The investigators will recruit a total of 200 patients with an eating disorder in the university hospital of Montpellier.

Participation consists of a one-day visit with a multidisciplinary assessment. No action is specific to research. This is the usual management of patients with eating disorders addressed to our department.

ELIGIBILITY:
Inclusion criteria :

* Patient with an eating disorder according to DSM-V criteria
* Patient aged from 15 to 65 years
* Patient who performs the day-hospital evaluation
* Patient affiliated to a French social security system
* Patient able to understand the nature, the aim and the methodology of the study For minor one of the legal guardians gave his consent

Exclusion criteria:

* Patient in an unstable somatic state (eg severe metabolic disorder making impossible or unreliable neuropsychological assessments)
* Patient's refusal to participate
* Patient protected by law (guardianship or curatorship)
* Pregnant or nursing women. A dosage of βHCG will be performed to ensure the absence of pregnancy.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with eating disorder
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Level of functional impairment assessed by the clinician with the FAST scale | 1 day
  We aim to investigate the link between global functioning and decision making abnormalities of patients with eating disorder.
  The Functioning Assessment Short Test (FAST) is composed of 24 items assessing various dimensions of daily functionning. Each item is ranged from 0 (no difficulty) to 3 (major difficulty) like a likert scale. The FAST is subdivided in 6 subscales : Autonomy (from 0 to 12), Professional activity (from 0 to 15), Cognitive functioning (from 0 to 15), Finances (from 0 to 6), interpersonal relationships (from 0 to 18) and Hobbies (from 0 to 6). The total score is the sum of the 6 subscales from 0 to 72. A hight score reveal hight difficulties in daily functionning

SECONDARY OUTCOMES:
Decision making assessed by the Iowa Gambling Task | 1 day
  We aim to investigate the link between decision making abnormalities and eating disorder caracteristicus
Level of cognitive flexibility assessed by the Brixton test | 1 day
  We aim to investigate the link between cognitive flexibility abnormalities and eating disorder caracteristicus
Level of central coherence assessed by the Rey Figure Test | 1 day
  We aim to investigate the link between central coherence abnormalities and eating disorder caracteristicus

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Guillaume, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC